CLINICAL TRIAL: NCT01516814
Title: Randomized, Open-label, Parallel-group, Active-controlled Study of Rivaroxaban in Patients With Acute Symptomatic Pulmonary Embolism, With or Without Symptomatic Deep Vein Thrombosis
Brief Title: Venous Thromboembolism (VTE) Treatment Study in Japanese Pulmonary Embolism (PE) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15960
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Embolism
Keywords: acute symptomatic pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Rivaroxaban; Heparin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 2 (Active Comparator)
  Interventions: Drug: Unfractionated heparin
- Arm 3 (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 15 mg twice daily for 21 days, followed by 15 mg once daily
  Arms: Arm 1
Drug: Unfractionated heparin — To be adjusted to maintain the activated partial thromboplastin time (aPTT) prolongation (1.5 to 2.5 times the control)
  Arms: Arm 2
Drug: Warfarin — To be adjusted on the basis of prothrombin time-international normalized ratio (PT-INR) values target range (1.5 to 2.5)
  Arms: Arm 3

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of rivaroxaban in the treatment of pulmonary embolism (PE) and the prevention of the occurrence and the recurrence of deep vein thrombosis (DVT) or PE in Japanese patients with acute symptomatic PE with or without symptomatic DVT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >/= 20 years of age in patients with confirmed acute symptomatic pulmonary embolism (PE) with or without symptomatic deep vein thrombosis (DVT)

Exclusion Criteria:

* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of PE
* More than 48 hours pre-randomization treatment with therapeutic dosages of anti-coagulant treatment or more than a single dose of warfarin from the onset of the current episode of PE to randomization
* Calculated creatinine clearance (CLCR) < 30 mL/min
* Subjects with hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk
* Active bleeding or high risk for bleeding contraindicating treatment with unfractioned Heparin (UFH) or warfarin
* Systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with newly onset of symptomatic venous thromboembolism (VTE) | Up to 12 months
Number of clinically relevant bleedings | Up to 2 days after last dose

SECONDARY OUTCOMES:
Number of participants with improvement in thrombotic burden | At week 3
Number of participants with deterioration in thrombotic burden | Up to 12 months
Number of participants with the composite of newly onset of symptomatic VTE or asymptomatic deterioration of thrombus | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- Japan (28):
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Aomori, Aomori
  - Chiba, Chiba
  - Sakura, Chiba
  - Kurume, Fukuoka
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Kahoku-gun, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Tsu, Mie-ken
  - Matsumoto, Nagano
  - Suwa, Nagano
  - Niigata, Niigata
  - Osaka, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Saga, Saga-ken
  - Shizuoka, Shizuoka
  - Shimotsuke, Tochigi
  - Bunkyo-ku, Tokyo
  - Chuoku, Tokyo
  - Itabashi-ku, Tokyo
  - Meguro-ku, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Matsuo H, Prins M, Lensing AW, Fujinuma EW, Miyamoto Y, Kajikawa M. Shortened length of hospital stay with rivaroxaban in patients with symptomatic venous thromboembolism in Japan: the J-EINSTEIN pulmonary embolism and deep vein thrombosis program. Curr Med Res Opin. 2015 Jun;31(6):1057-61. doi: 10.1185/03007995.2015.1037728. Epub 2015 May 11. PMID 25851062
- [Derived] Yamada N, Hirayama A, Maeda H, Sakagami S, Shikata H, Prins MH, Lensing AW, Kato M, Onuma J, Miyamoto Y, Iekushi K, Kajikawa M. Oral rivaroxaban for Japanese patients with symptomatic venous thromboembolism - the J-EINSTEIN DVT and PE program. Thromb J. 2015 Jan 17;13:2. doi: 10.1186/s12959-015-0035-3. eCollection 2015. PMID 25717286